CLINICAL TRIAL: NCT00051961
Title: Effects of Dopaminergic Agonist Treatment on Spinal Cord Excitability in Restless Legs Syndrome
Brief Title: Effect of Ropinirole on Spinal Cord Reflexes and Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030075; 03-N-0075
Record Dates: First submitted 2003-01-17; First posted 2003-01-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-18

CONDITIONS: Restless Legs Syndrome
Keywords: Dopamine; Spinal Physiology; Flexor Reflex; Ropinirole; Motor Control; Dopaminergic; Restless Legs
MeSH Terms: conditions — Restless Legs Syndrome

SUMMARY:
This study will examine the effects of the drug Ropinirole on spinal cord reflexes and on symptoms of restless legs syndrome (RLS). Patients with RLS have uncomfortable sensations in the legs, usually in the evening or early part of the night. Most patients also have periodic involuntary leg movements. The condition tends to worsen over time, resulting in severe discomfort and sleep disturbances. Ropinirole affects chemical messengers thought to be involved in spinal cord function and in modulating RLS symptoms.

Healthy normal volunteers and patients with RLS between 18 and 80 years of age may be eligible for this study. Patients must have mild to moderate RLS and periodic limb movements. All candidates will be screened with a medical history, physical and neurological evaluations, electromyogram (see below), polysomnogram (see below), electrocardiogram (ECG), and blood and urine tests. They may also have magnetic resonance imaging (MRI) or computerized tomography (CT) scans and a chest x-ray. Participants must stop taking all medications prohibited by the study for at least 1 week before the study starts and throughout its duration.

The study will last approximately 2 to 3 weeks for healthy volunteers and 7 to 8 weeks for patients. Participants will undergo the following baseline evaluations: electroencephalography (EEG), a measure of brain wave activity; polysomnography (PSG), an overnight sleep study; electromyography (EMG), a measure of muscle activity; and spinal flexor reflex studies (spinal cord responses to electrical stimulation). For these studies, several electrodes are attached to the scalp or to the legs and arms using a cream that helps conduct brain signals through the cables to be recorded. The nervous system activity can be assessed at rest or after stimulation with an electric current. For EMG, a small needle is inserted into a few muscles and the subject is asked to relax or to contract the muscles. The electrical activity of the muscle cells is recorded and analyzed by a computer. Spinal flexor reflex studies usually involve stimulating the nerves in the legs with very brief electric currents of mild to moderate intensity. Flexor reflex studies will be done early in the night while the subject is awake and also during sleep. Brain, muscle and breathing activities will be monitored continuously during sleep.

A suggested immobilization test (SIT) will be done around 10 p.m. During the test, the subject sits still for about 1 hour, while the leg muscle activity is recorded using special electronic devices attached to the skin. At the end of the test, volunteers will be asked questions about symptoms they may have experienced during the test, and patients will be asked questions about their RLS symptoms during the test.

After the baseline tests, participants will be randomly assigned to take either Ropinirole tablets or a placebo (a look-alike inactive substance) daily for 5 weeks. They will be admitted to the NIH Clinical Center for 3 to 4 nights at the end of the second week and for 2 nights at the end of the study to repeat the baseline tests described above. Volunteers will take Ropinirole or placebo daily for 1 week. They will be admitted to the Clinical Center for 3 to 4 days at the beginning and then at the end of the study for repeat testing.

Medical examinations, ECGs and blood tests will be done at various times during the study for safety monitoring. Patients' blood pressure will be monitored weekly. Small amounts of blood will be drawn up to three times each day for routine studies, research and drug levels. Throughout the study volunteers will complete questionnaires for evaluation of possible RLS symptoms, and patients will have their symptoms assessed using a RLS Severity Rating Scale. Two weeks after the study ends, participants will be interviewed by telephone about any adverse experiences.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of stimulation of dopaminergic D2, D3 receptors on spinal cord excitability and on the severity of symptoms in patients with mild to moderately advanced restless legs syndrome. In a controlled proof-of-principle clinical study, the acute efficacy of ropinirole will be assessed through the use of validated electrophysiological tests and severity scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who meet all of the following inclusion criteria at screening or Day 0 will be eligible to participate in the study:

1. Male or female subjects aged 18 to 80.
2. Body Mass Index within the range 19-34 kg/m(2) inclusive.
3. For patients only, diagnosed with mild to moderate RLS based on the presence of a characteristic clinical history and the IRLSSG diagnostic criteria.
4. Normal physical and neurological examination.
5. Subject is willing to adhere to protocol requirements as evidenced by written, informed consent.
6. No clinical significant abnormalities on clinical chemistry or haematology examination at the pre-study medical evaluation.
7. A normal 12 lead ECG at the pre-study medical.
8. A negative pre-study Hepatitis B surface antigen and Hepatitis C antibody result within 3 months of the start of the study.
9. Negative pre-study urine drug screen.
10. RLS Rating Scale score of greater than or equal to 15 at the time of baseline evaluation, after medication wash out.
11. Presence of PLMs by convincing history, or document by SIT or polysomnography tests at the time of baseline evaluation.

EXCLUSION CRITERIA:

Subjects meeting any of the following exclusion criteria either at Day 0 or during the study will not be enrolled or will be immediately excluded from the study, as appropriate:

1. History of any medical condition that can reasonably be expected to subject the individual to unwarranted risk or compromise scientific integrity of the study;
2. History or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion drugs
3. Clinically significant laboratory abnormalities including liver enzyme elevation greater than twice the upper limit of normal;
4. Patient unwilling or unable to stop their usual medications for RLS;
5. Subjects unable or unwilling to discontinue a prohibited concomitant medication;
6. Subjects who have received prescribed medication within 7 days prior to the first dosing day (defined as Day 1), which in the opinion of the Principal Investigator will interfere with the study procedures or compromise safety.
7. Withdrawal, introduction, or change in dose of hormone replacement therapy (HRT) and/or any drug known to substantially inhibit or induce CYP1A2 within 2 weeks prior to first dose (Day 1).
8. Patients suffering from RLS symptoms during the daytime (daytime defined as 10.00 until 16.00 hours).
9. Subjects who have not been using a clinically accepted contraceptive method (such as oral contraception, surgical sterilization, IUD, diaphragm in conjunction with spermicidal foam and condom on the male partner, or systemic contraception) for the last 30 days, or is not at least one year post-menopausal (if female);
10. Subjects who are pregnant or breastfeeding;
11. Subjects with cognitive impairment (MMSE less than 25);
12. Subjects who have participated in a clinical study with an investigational drug within the last 3 months;
13. Subjects with history or presence of active drug or alcohol abuse that, in the opinion of the investigators, would interfere with compliance or safety or scientific integrity of study;
14. Subjects unwilling to sign an informed consent or to comply with protocol requirements.
15. A dissomnia or parasomnia other than, in patients, primary RLS (e.g. narcolepsy, sleep tenor disorder, sleepwalking disorder, and breathing-related sleep disorder), either from clinical review or from polysomnography (including subjects with apnea hypopnea index greather than 5/h).
16. Signs of secondary RLS (e.g. renal failure (end-stage renal disease), iron deficient anemia or pregnancy at baseline).
17. Subjects with clinical and/or biochemical evidence of iron deficiency.
18. Subjects with a diastolic blood pressure greater than or equal to 110mmHg or less than or equal to 50mmHg OR systolic blood pressure greater than or equal 180mmHg or less than or equal 90mmHg at baseline.
19. Subjects with known intolerance to ropinirole or other dopaminergic agonist.
20. Patients with symptomatic orthostatic hypotension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-01-14; Study Completion 2007-10-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Trenkwalder C, Hening WA, Walters AS, Campbell SS, Rahman K, Chokroverty S. Circadian rhythm of periodic limb movements and sensory symptoms of restless legs syndrome. Mov Disord. 1999 Jan;14(1):102-10. doi: 10.1002/1531-8257(199901)14:13.0.co;2-e. PMID 9918351